CLINICAL TRIAL: NCT00001346
Title: Diabetic Retinopathy and Visual Function Study
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930037; 93-EI-0037
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Diabetic Retinopathy; Macular Degeneration; Vision, Subnormal
Keywords: Diabetic Macular Edema; Diabetic Retinopathy; Macular Edema; Photocoagulation; Psychophysical Testing; Stiles-Crawford Effect
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Vision, Low; Macular Edema

SUMMARY:
The purpose of this study is to evaluate possible mechanisms of central visual loss in patients with diabetes mellitus. The visual loss of interest to be investigated is that associated with macular edema (prior to and following laser photocoagulation treatment) and that associated with panretinal photocoagulation. The evaluation will be performed with psychophysical testing, i.e., static perimetry and contrast sensitivity function. Of particular interest, the mechanisms of visual loss associated with macular edema (prior to and following laser photocoagulation) will be further investigated. Photoreceptor-mediated visual loss will be assessed by measurements of the Stiles-Crawford effect. Visual loss mediated by post-receptoral retinal changes will be assessed by measuring the Westheimer spatial desensitization/sensitization effect.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate possible mechanisms of central visual loss in patients with diabetes mellitus. The visual loss of interest to be investigated is that associated with macular edema (prior to and following laser photocoagulation treatment) and that associated with panretinal photocoagulation. The evaluation will be performed with psychophysical testing, i.e., static perimetry and contrast sensitivity function. Of particular interest, the mechanisms of visual loss associated with macular edema (prior to and following laser photocoagulation) will be further investigated. Photoreceptor-mediated visual loss will be assessed by measurements of the Stiles-Crawford effect. Visual loss mediated by post-receptoral retinal changes will be assessed by measuring the Westheimer spatial desensitization/sensitization effect.

ELIGIBILITY:
Patients with diabetic retinopathy that has not been previously treated are eligible for the study.

Patients who have had laser photocoagulation (either focal or scatter) are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1992-11; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Higgins KE, Meyers SM, Jaffe MJ, Roy MS, de Monasterio FM. Temporary loss of foveal contrast sensitivity associated with panretinal photocoagulation. Arch Ophthalmol. 1986 Jul;104(7):997-1003. doi: 10.1001/archopht.1986.01050190055039. PMID 3729795
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. II. Prevalence and risk of diabetic retinopathy when age at diagnosis is less than 30 years. Arch Ophthalmol. 1984 Apr;102(4):520-6. doi: 10.1001/archopht.1984.01040030398010. PMID 6367724
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. III. Prevalence and risk of diabetic retinopathy when age at diagnosis is 30 or more years. Arch Ophthalmol. 1984 Apr;102(4):527-32. doi: 10.1001/archopht.1984.01040030405011. PMID 6367725